CLINICAL TRIAL: NCT04395742
Title: 1,3,7-Trimethylxanthine as a Treatment of COVID-19: Results of a Controlled Study
Acronym: TMX COVID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TMX COVID
Record Dates: First submitted 2020-05-14; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coffee:1,3,7-trimethylxanthine
  Interventions: Other: Data collection
- Tea and hot chocolate with milk
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Only data collection

SUMMARY:
This is observational study to assess the prognosis of patients hospitalized with COVID-19 confirmed by RT-PCR and exposed to trimethylxanthine (TMX).

Trimethylxanthine is the active molecule present in coffee. Due to the lack of etiologic treatments and considering interest about old treatments as an avenue for research, we conducted a comparative study aiming to evaluate the effect of 1,3,7-trimethylxanthine on COVID-19 infected patients. This is actually a study about methodology.

The objective of this study is therefore not to demonstrate the effect of the substance on the disease but the importance of a rigorous methodology in scientific research. This project is called "Method and Teaching of Scientific Studies".

ELIGIBILITY:
Inclusion Criteria:

* Age > 18,
* No Trimethylxanthine contraindications (defined as allergy, previous reported secondary effects),
* Infectious Disease Unit admission.

Exclusion Criteria:

* Secondary effects about Trimethylxanthine,
* Refuse to participate

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients meeting the eligibility criteria and wishing to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of vital status | 6 days
  the patient clinical status at day 6 after hospital admission, defined as alive, or dead.

SECONDARY OUTCOMES:
Comparaison of duration of hospital stay | 6 days
Comparaison of severity | 6 days
  Evaluated by National Early Warning Score from 0 to 20, 20 being the worst score, with a high risk of death.
Comparaison of secondary effects (adverse events that needed disruption of treatment (anemia, tachycardia, osteoporosis) : secondary effects of coffee). | 6 days
  with
Comparaison of use of antibiotics | 14 days after hospital admission.

REFERENCES:
- [Derived] Belaroussi Y, Roblot P, Peiffer-Smadja N, Delaye T, Mathoulin-Pelissier S, Lemeux J, Le Moal G, Caumes E, Roblot F, Bleibtreu A. Why Methodology Is Important: Coffee as a Candidate Treatment for COVID-19? J Clin Med. 2020 Nov 17;9(11):3691. doi: 10.3390/jcm9113691. PMID 33213035